CLINICAL TRIAL: NCT05481723
Title: Lung Ultrasound-guided Hemodynamic Optimization in Major Non-cardiac Surgery: a Randomized Control
Brief Title: Lung Ultrasound-guided Hemodynamic Optimization
Acronym: POINTBAR
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Centre Hospitalier Universitaire, Amiens (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: PI2021_843_0081
Record Dates: First submitted 2022-07-28; First posted 2022-08-01 (Actual); Last update posted 2025-05-28 (Actual); Status verified 2025-05

CONDITIONS: Lung Ultrasound; Goal Directed Therapy; Non-cardiac Surgery
Keywords: lung ultrasound; goal directed therapy; non-cardiac surgery
MeSH Terms: interventions — Norepinephrine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Control group (Active Comparator): The control group will be treated according to the usual protocol of the department (standard group)
  Interventions: Drug: noradrenaline and vascular filling
- pulmonary ultrasound group (Experimental): the experimental group follows an algorithm incorporating the number of B-lines occurring after a filling test (pulmonary ultrasound group).
  Interventions: Procedure: pulmonary ultrasound after vascular filling

INTERVENTIONS:
Drug: noradrenaline and vascular filling — In the control group, the haemodynamic management of the patients is done according to usual practice by maintaining blood pressure with noradrenaline and optimising stroke volume with vascular filling.
  Arms: Control group
Procedure: pulmonary ultrasound after vascular filling — In the interventional group, intraoperative haemodynamic management is based on an algorithm that includes measurement of the number of B-lines appearing on pulmonary ultrasound after vascular filling. Monitoring of the stroke volume will also be performed in this group in order to stop the vascular filling if the ESV does not increase by more than 10%.
  Arms: pulmonary ultrasound group

SUMMARY:
The formalized expert recommendation of the French Society of Anesthesia and Intensive Care recommends guiding vascular filling by measuring the stroke volume (SV) in surgical patients considered at high risk. Vascular filling should be continued in the event of preload dependence and stopped in the event of the appearance of preload independence. The aim is to avoid vascular overload due to excessive vascular filling. The application of this recommendation has resulted in a reduction in postoperative morbidity, length of hospital stay and time to return to oral feeding. The superiority of this strategy is now being questioned and the predictive indices of response to vascular filling (static and dynamic) have many limitations. In addition, none of the cardiac output monitors are the gold standard for intraoperative use.

Through the study of artefacts, lung ultrasound has been gaining ground over the last twenty years, particularly in cardiology, nephrology and intensive care. By analogy with radiological B-lines, ultrasound B-lines result from the reverberation of ultrasound on the subpleural inter-lobular septa thickened by oedema. The Fluid Administration Limited by Lung Sonography (FALLS) protocol, described by Lichtenstein et al, is defined as the visualisation of new B lines during a vascular filling test. If a B-line appears in an area where it was not present during vascular filling, the most likely diagnosis is hydrostatic overload of the subpleural interstitial septum. This appearance of B-lines occurs at a sub-clinical stage.

The use of lung ultrasound could allow real-time assessment of vascular filling and its tolerance during the intraoperative period. The main objective of the study is to demonstrate a decrease in the incidence of postoperative complications (organ failure) (as defined by international guidelines) when using lung ultrasound-guided haemodynamic optimisation compared to standard optimisation.

ELIGIBILITY:
Inclusion Criteria:

* Age> 18 years old
* Abdominal, orthopaedic or vascular surgery with general anaesthesia
* Patient of legal age ≥ 18 years.
* ASA score ≥ II
* Estimated duration of surgery > 2 hours
* At least two of the following comorbidities (age > 50 years, hypertension, heart disease, electrocardiogram (ECG) abnormality, acute pulmonary oedema, smoking, stroke, peripheral arterial disease, non-insulin dependent or insulin dependent diabetes, ascites, chronic renal failure)
* Signed consent.
* Affiliation to a social security scheme.

Exclusion Criteria:

* Severe untreated or unbalanced hypertension on treatment.
* Preoperative renal failure on dialysis.
* Acute heart failure.
* Acute coronary insufficiency.
* Vascular surgery with renal plasty.
* Cardiac surgery.
* Preoperative shock.
* Refusal of patient participation.
* Pregnant, parturient or breastfeeding woman.
* Patient under guardianship or private law.
* Acute respiratory distress syndrome according to the Berlin definition
* respiratory distress not fully explained by cardiac failure or increased blood volume,
* PaO2/FiO2 ratio ≤ 300 mm Hg on mechanical ventilation (invasive or non-invasive)
* Chronic respiratory failure with home oxygen therapy.
* Chronic interstitial lung disease
* Presence of an acoustic barrier (pneumothorax, subcutaneous emphysema, pleural calcifications, chest bandage, gunshot shrapnel...)
* Participation in other interventional drug research.
* Surgical fields covering the sites of investigation in lung ultrasound.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 350 (Estimated)
Dates: Start 2022-07-28 (Actual); Primary Completion 2027-07 (Estimated); Study Completion 2027-08 (Estimated)

PRIMARY OUTCOMES:
Number of Postoperative Organ failure | within 7 days
  Organ failure is defined according to the recommendations of the European Society of Anaesthesia (ESA)

SECONDARY OUTCOMES:
length of hospital stay | 7 days
  Number of days staying in hospital

CONTACTS AND LOCATIONS:
Locations (1):
- CHU Amiens, Amiens, France

IPD SHARING:
Plan to Share IPD: No